CLINICAL TRIAL: NCT01870154
Title: Effectiveness of an Intervention for Prevention and Treatment of Burnout in Primary Health Care Professionals
Brief Title: Effectiveness of an Intervention for Prevention and Treatment of Burnout in Primary Care
Acronym: EDESPROAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 08/1443
Record Dates: First submitted 2013-06-02; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Burnout Syndrome
Keywords: Burnout syndrome; Job stressors; Primary Health Care; Health professional
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention consists of 16 hours of training, to be held at the subject's health center. The workshop involves mixed learning, comprising 4 sessions, each 2 hours long, in addition to personal work previous to and after each session of reading relevant bibliography and performing exercises, self-evaluation, and case studies (8 hours of individual work).
  Interventions: Behavioral: Training
- Control group (Active Comparator): Usual care
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — The objective of the intervention is learning from the work experience of professionals attending the workshop to know and recognize the risk and process of the burnout syndrome and the characteristics specific to the health setting, as well as promoting prevention lines by transmitting strategies to manage and control the elements and consequences of the syndrome process (physical, psychological, and social).

SUMMARY:
Background: Burnout syndrome is an important health problem that affects many professionals and must be addressed globally, with both organizational measures and personal interventions. Burnout of health professionals can be prevented in order to avoid personal, familial, and social consequences, as well as repercussions for patients.

Methods/Design: This work describes a protocol for a controlled, pragmatic, randomized clinical trial in 2 parallel groups: intervention and control. All health professionals from 7 health care centers (HCCs) will form the intervention group, and all health professionals from 7 different HCCs will form the control group. The intervention group will receive 16 hours of training at their work place. The Maslach's burnout inventory (MBI), burnout physician Questionnaire (CDPM) or burnout nurse Questionnaire (CDPE), and the 28-item Goldberg's General Health Questionnaire (GHQ-28), validated for our setting, will be used as measurement tools. Change in the average scores from the MBI emotional exhaustion scale will be compared between the intervention and control groups, measured as intention-to-treat, and the intervention will be considered effective if a minimum increase of 20% is achieved.

Discussion: Due to the deleterious consequences of burnout syndrome for people suffering from it and for the organization where they work, it is necessary to evaluate the effectiveness of certain interventions for its prevention. Organizational measures are important for preventing burnout syndrome, but so is providing professionals with coping strategies, as this group intervention intends to do.

ELIGIBILITY:
Inclusion Criteria:

* All health professionals (family physicians, pediatricians, and nurses) who are part of the health care centers at the moment of the trial.

Exclusion Criteria:

* No one.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maslach's burnout inventory (MBI) | One year
  Worker classification regarding burnout syndrome will be performed according to the MBI, which includes 22 items to evaluate emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF), with scores ranging from 0 to 6 on the Likert scale. We consider a high degree of burnout in the case of EE ≥ 27 points, DP ≥ 10, and PF <33. Moderate burnout will be considered in the case of 26<EE<19 points, 6<DP<9 points, and 34<PF<39 points. Low levels will be considered for EE≤18 points, DP≤5 points, and PF≥40 points.

SECONDARY OUTCOMES:
Goldberg's General Health Questionnaire (GHQ-28) | One year
  It consists of 28 items, divided into 4 sub-scales. It is used to estimate the prevalence of psychiatric disease in a specific population and discover cases of psychiatric pathologies in non specialized consultations. It is not appropriate for performing clinical diagnosis, but can be employed to evaluate symptomatology using its sub-scales: A (somatic symptoms), B (anxiety/insomnia), C (social dysfunction), and D (severe depression). There are 4 possible answers to each question. The Likert scoring system assigns a value from 0 to 3 to each of the 4 possible answers.

CONTACTS AND LOCATIONS:
Overall Officials: Tomás Gómez-Gascón, MD, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (1):
- Gerencia de Atención Primaria, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Gomez-Gascon T, Martin-Fernandez J, Galvez-Herrer M, Tapias-Merino E, Beamud-Lagos M, Mingote-Adan JC; Grupo EDESPROAP-Madrid. Effectiveness of an intervention for prevention and treatment of burnout in primary health care professionals. BMC Fam Pract. 2013 Nov 17;14:173. doi: 10.1186/1471-2296-14-173. PMID 24237937